CLINICAL TRIAL: NCT06876935
Title: Guac & Grow: Early Avocado Exposure on Development and the Gut Microbiome in American Hispanic Infants
Brief Title: Early Avocado Exposure on Development and the Gut Microbiome in American Hispanic Infants
Acronym: Guac & Grow
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Corrie Whisner, Associate Professor, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00021667; AWD00040492 (Other Grant/Funding Number: Avocado Nutrition Center)
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Gut Microbiome; Neurocognitive Correlates of Eating Habits; Infant Growth
Keywords: avocado; infants; complimentary feeding; growth; development; gut microbiome; neurocognitive; brain health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily Avocado (Experimental): Infants in the daily avocado group will receive a daily exposure amount of avocado ranging from 1/4 (~37.5 g or 1.25 oz) to 1/2 (~75 g or 2.5 oz) of a medium-sized avocado.
  Interventions: Other: Daily avocado
- No Avocado Control (No Intervention): Infants in the control group will be asked to limit avocado exposure to no more than 1/8 of a medium-sized avocado (~19 g, 2 Tbs) once per week.

INTERVENTIONS:
Other: Daily avocado — Infants in the daily avocado group will receive a daily exposure amount of avocado ranging from 1/4 (~37.5 g or 1.25 oz) to 1/2 (~75 g or 2.5 oz) of a medium-sized avocado. At 6-8 months, infants will be provided 1/4 (~37.5 g or 1.25 oz) of a medium-sized avocado for daily consumption. Then from 9-12 months, they will begin receiving 1/2 (~75 g or 2.5 oz) of a medium-sized avocado for daily consumption.
  Arms: Daily Avocado

SUMMARY:
The goal of this clinical trial is to learn if daily avocado intake can improve growth and brain and gut health in infants. The main questions it aims to answer are:

Does daily eating of avocados change which microbes live in the infant's gut? Does daily avocado intake improve infant motor skills and cognitive development?

Researchers will compare avocado intake to standard of care (no or limited avocado intake) to see if regular avocado intake from 6-12 months of life influences gut and brain health.

Participating mothers/guardians and their infants will:

Parents will provide avocado or no avocado to their infant every day for 6 months starting around 6 months of infant age.

Parents will allow study staff to visit participant homes to collect data via surveys and observations and measure infant growth.

Parents will swab soiled infant diapers for gut microbe measures. Parents will keep a diary of the infant's avocado consumption and acceptance of the food.

Parents will record their infant's dietary intake

DETAILED DESCRIPTION:
The overarching goal of this two-arm, randomized clinical trial, is to study how early avocado exposure impacts the gut microbiome and developmental milestones in Hispanic infants. The following aims will be achieved using a randomized, parallel-arm, clinical trial.

Specific Aim 1: Evaluate how avocado consumption modulates the infant GM. Hypothesis 1: Daily avocado exposure will produce distinct structural and functional signatures within the GM compared to control.

Specific Aim 2: Investigate how avocado consumption affects emerging motor and neurocognitive skills in infants.

Hypothesis 2: Daily avocado exposure will improve development compared to the control group.

All measures will be completed at participant homes when infants are 6, 9, and 12 months of age. Infants in the intervention arm will receive a daily amount of avocado and the amount consumed will be measured. Those in the control arm will be asked to limit avocado exposure to no more than once per week.

Those in the control arm will receive the same quantity of avocados for 6 months to provide to their child once the 6-month intervention period has been completed so that control infants may also benefit from avocado consumption.

ELIGIBILITY:
Inclusion Criteria:

* 4-6-month-old Hispanic/Latine, non-preterm (>37 weeks gestation) singleton infants
* Infants born to mothers 18 years and older while pregnant
* Parents speak English and/or Spanish
* Families willing to begin feeding infants avocado around 6 months of age or when the infant is ready for solids for a total of 6 months
* Family history of food or latex allergies will be evaluated as avocado is a latex fruit and can cause allergic responses. If either mom or dad is allergic to avocado, physician clearance for infant participation will be needed.
* At least one caregiver in the home must have at least an 8th-grade education level

Exclusion Criteria:

* Infants with growth, chromosomal, or genetic abnormality, developmental and cognitive impairments, or severe comorbidity that could impact growth and development
* Infants born with congenital abnormalities or developmental delays
* Infant birth weights <2500 g or >4000 g
* Infants introduced to solid foods prior to 3 months of age
* Biological mothers with known substance use during pregnancy (alcohol, tobacco, marijuana, or illegal drugs), or who experienced a high-risk pregnancy (e.g., preeclampsia, diabetes-Types 1 and 2 and gestational, HIV, etc.)

Ages: 3 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome | At enrollment to the end of treatment at 6 months
  Parents will collect stool samples from infant diapers using sterile swabs (parent will swab a soiled diaper) and backup soiled diapers.

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scale (Vinland-3) | From enrollment to the end of treatment at 6 months
  A questionnaire completed by the parent/caregiver that is normed for ages from birth through 90 years. The tool assesses adaptive behaviors (things people do to function in everyday life) in three domains: communication, daily living skills, and socialization.
McArthur Bates Communicative Development Inventories III (MBCDI-III) | From enrollment to the end of treatment at 6 months
  A widely used checklist completed by parents to assess children's early communication skills such as comprehension and use of gestures and words.
HOME Assessment | From enrollment to the end of treatment at 6 months
  Research personnel will objectively evaluate the caring environment in which a child is raised and parent-child interaction using this validated assessment.
Mullen Scales of Early Learning | From enrollment to the end of treatment at 6 months
  Study staff will administer a structured 15-minute play session with the infant to objectively assess motor, visual, and early language skills.
Infant length | From enrollment to the end of treatment at 6 months
  Infant length will be assessed with a pediatric length board and reported in centimeters.
Infant weight | From enrollment to the end of treatment at 6 months
  Infant weight will be assessed with a calibrated scale and reported in grams.

OTHER OUTCOMES:
Skin Carotenoid Concentration | From enrollment to the end of treatment at 6 months
  The Veggie-Meter, a non-invasive measurement device, will be used to assess the carotenoid content on the index finger of the infant's right hand using reflection spectroscopy via a 2 mm wide white LED light (similar to pulse oximeter measures on the index finger).
Infant 24-hour Diet Records | From enrollment to the end of treatment at 6 months
  Habitual intake will be assessed via the Automated Self-Administered 24-hr recall software (ASA24) on 2 weekdays and one weekend day developed by the National Cancer Institute.
Food intake photos | From enrollment to the end of treatment at 6 months
  Pre-post meal photos of the infant and their food will be provided by the parents. These images will be used to help corroborate dietary intake and behavior data.
Centers for Disease Control Infant Feeding Practices Study II Questionnaire | From enrollment to the end of treatment at 6 months
  This questionnaire asks about breastfeeding, formula feeding, complementary feeding, introduction to solid foods, food allergies, and participation in the Special Supplemental Nutrition Assistance Program for Women, Infant, and Children.
Food Security Screener | From enrollment to the end of treatment at 6 months
  The USDA 6-Item Food Security Screener will be used to assess household food insecurity.
Stool Consistency | From enrollment to the end of treatment at 6 months
  Parents will be asked to classify the stool consistency using the picture-based Brussels Infant and Toddler Stool Scale (BITSS), developed specifically for non-toilet-trained children.

CONTACTS AND LOCATIONS:
Overall Officials: Corrie M Whisner, PhD, Principal Investigator — Arizona State University
Locations (1):
- College of Health Solutions, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
To comply with the rigor and reproducibility goals of the scientific community, we will make data available when required for publication in peer-reviewed scholarly journals. Any data shared for publication will be shared in repositories such as those managed by the U.S. government (e.g. dbGAP for microbiome sequence files and associated phenotype metadata) or Arizona State University. Data will be shared with the sponsor and made available for secondary data analyses upon reasonable investigator request. Further study protocols will be made available upon request to the PI and analytical code and statistical analyses will be shared through GitHub.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting information will be available no earlier than the time of first publication.
Access Criteria: IPD will be accessible to investigators interested in engaging in secondary data analysis or recreating analyses done by the study team as educational exercises.